CLINICAL TRIAL: NCT02464488
Title: Study of Interindividual Variability in the Response to New Oral Direct Anticoagulants (Dabigatran Etexilate, Rivaroxaban or Apixaban) in Patients 80 Years Old and Over, Using a Population Pharmacokinetics Approach.
Brief Title: New Oral Direct Anticoagulants in Patients 80 Years Old and Over : a Population Pharmacokinetics Study
Acronym: ADAGE
Status: Completed | Type: Observational
Sponsor: Hôpital Charles Foix (Other)
Collaborators: University of Paris 5 - Rene Descartes (Other); Sorbonne University (Other); Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: cfx-adage-2015
Record Dates: First submitted 2015-06-02; First posted 2015-06-08 (Estimated); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Atrial Fibrillation
Keywords: Anticoagulants; Factor Xa Inhibitors; Antithrombins; Pharmacokinetics; Aged, 80 years and older
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Main cohort (only cohort of the study): Patients aged 80 years or older under treatment with dabigatran, rivaroxaban or apixaban because atrial fibrillation. All patients will have plasma drug concentrations measured and will be followed afterwards similarly
  Interventions: Other: Plasma drug concentrations

INTERVENTIONS:
Other: Plasma drug concentrations — Measure of plasma concentrations of the anticoagulant drug taken by the patient

SUMMARY:
Several new oral direct anticoagulants have been recently marketed. However, only a few, limited, studies have provided data about the pharmacology of new oral direct anticoagulants in older persons. This study try to better define wether the pharmacology of each of these 3 drugs (dabigatran, rivaroxaban and apixaban) is actually significantly different in very older patients (over 80) and to which extend. The investigators also try to characterize the main determinants (age, weight, renal function, co-morbidities, etc) of the variability observed between individuals in their response to he drugs studied. The method employed is a population pharmacokinetic/pharmacodynamic study.

DETAILED DESCRIPTION:
Several new oral direct anticoagulants have been recently marketed. A main indication for taking these drugs is atrial fibrillation and, in everyday practice, most patients with atrial fibrillation are older people. However, only a few, limited, studies have provided data about the pharmacology of new oral direct anticoagulants in older persons. Furthermore, this limited data strongly suggests that, in older patients, mean concentrations, overall exposition and half-live of these drugs are increased, as compared with younger people. This study try to better define wether the pharmacology of each of these 3 drugs (dabigatran, rivaroxaban and apixaban) is actually significantly different in very older patients (over 80) and to which extend. The investigators also try to characterize the main determinants (age, weight, renal function, co-morbidities, etc) of the variability observed between individuals in their response to he drugs studied. The method employed is a population pharmacokinetic/pharmacodynamic study. This is, many people (projected 225 patients) will have a few blood samples each and all data will be pooled using statistical methods specific to this kind of studies. Each patient will have one to five blood samples, taken at te same time that routine blood analysis, to determine plasma concentrations of the studied drug. In addition, patients will be followed for thrombotic and haemorrhagic events at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 80 years or older
* Under treatment with dabigatran, rivaroxaban or apixaban
* For non-valvular atrial fibrillation

Exclusion Criteria:

* Mechanical (non-biological) heart valve
* Any severe condition leading to a short estimated life expectance (a few months)

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 80 years or older under treatment with dabigatran, rivaroxaban or apixaban because atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-08-25 (Actual)

PRIMARY OUTCOMES:
Pharmacologic parameters of new oral anticoagulants in elderly patients | 1 to 3 weeks
  Estimated area under the curve (AUC) of each of the 3 drugs studied

SECONDARY OUTCOMES:
Thromboembolic events | 1 year
  Any thromboembolic event (composite of ischemic stroke, systemic embolism or acute coronary syndrome) in the year after inclusion
Hemorrhagic events | 1 year
  Major hemorrhagic events in the year after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Carmelo Lafuente, MD, PhD, Principal Investigator — Hôpital Charles Foix, APHP, Université Paris 6 UPMC; Julien Le Guen, MD, Principal Investigator — Hôpital Européen Georges Pompidou, APHP, Université Paris 5 Descartes
Locations (2):
- France (2):
  - Hôpital Charles Foix, Ivry-sur-Seine, Île-de-France Region
  - Hôpital Européen Georges Pompidou, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No